CLINICAL TRIAL: NCT04116437
Title: A Phase 2, Multicenter, Single-arm Study of Zanubrutinib (BGB-3111) in Patients With Previously Treated B-Cell Lymphoma Intolerant of Prior Treatment With Ibrutinib and/or Acalabrutinib
Brief Title: Zanubrutinib (BGB-3111) in Participants With Previously Treated B-Cell Lymphoma Intolerant of Prior Bruton Tyrosine Kinase Inhibitor (BTKi) Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-215
Expanded Access: NCT04052854 (No longer available)
Record Dates: First submitted 2019-10-01; First posted 2019-10-04 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Waldenstrom Macroglobulinemia
Keywords: BGB-3111; Zanubrutinib; Ibrutinib Intolerance; BTK Inhibitor; Acalabrutinib Intolerance
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib (Experimental): Cohort 1: Chronic lymphocytic leukemia (CLL)/ small lymphocytic lymphoma (SLL), Waldenström macroglobulinemia (WM), mantle cell lymphoma (MCL), or marginal zone lymphoma (MZL) previously treated with ibrutinib
  Cohort 2: Chronic lymphocytic leukemia (CLL)/ small lymphocytic lymphoma (SLL), Waldenström macroglobulinemia (WM), mantle cell lymphoma (MCL), or marginal zone lymphoma (MZL) previously treated with acalabrutinib alone/with ibrutinib
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Zanubrutinib (BGB-3111) will be orally administered at a dose of 160 mg twice daily or 320mg once daily until disease progression, unacceptable toxicity, treatment consent withdrawal, or study termination.
  Other Names: BGB-3111; BRUKINSA

SUMMARY:
The primary objective of this study is to evaluate the safety of zanubrutinib (also known as BGB-3111) in chronic lymphocytic leukemia/small lymphocytic lymphoma, Waldenström macroglobulinemia, mantle cell lymphoma, or marginal zone lymphoma patients who have become intolerant of prior ibrutinib and/or acalabrutinib treatment, by comparing intolerance to adverse event profile as assessed by the recurrence and the change in severity of adverse events.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants must meet protocol defined disease criteria requiring treatment for their respective disease prior to initiation of ibrutinib or acalabrutinib
2. Ibrutinib and acalabrutinib intolerance is defined as an unacceptable toxicity where, in the opinion of the investigator, treatment should be discontinued in spite of optimal supportive care as a result of one of the following:

   1. For ibrutinib and acalabrutinib intolerance events:

      * 1 or more ≥ Grade 2 nonhematologic toxicities for >7 days (with or without treatment)
      * 1 or more ≥ Grade 3 nonhematologic toxicity of any duration
      * 1 or more Grade 3 neutropenia with infection or fever of any duration; or
      * Grade 4 heme toxicity which persists to the point that the investigator chose to stop therapy due to toxicity NOT progression.
   2. For acalabrutinib intolerance events only;

      * 1 or more ≥ Grade 1 nonhematologic toxicities of any duration with > 3 recurrent episodes; or
      * 1 or more ≥ Grade 1 nonhematologic toxicities for > 7 days (with or without treatment); or
      * Inability to use acid-reducing agents or anticoagulants (eg, proton pump inhibitors, warfarin) due to concurrent acalabrutinib use
3. Ibrutinib and/or acalabrutinib-related ≥ Grade 2 toxicities must have resolved to ≤ Grade 1 or baseline prior to initiating treatment with zanubrutinib. Grade 1 acalabrutinib-related toxicities must have resolved to Grade 0 or baseline prior to initiating treatment with zanubrutinib.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
5. Absolute neutrophil count (ANC) ≥ 1000/mm^3 with or without growth factor support and platelet count ≥ 50,000/mm^3 (may be post-transfusion), on or prior to C1D1 of zanubrutinib

Key Exclusion Criteria:

1. Clinically significant cardiovascular disease including the following:

   1. Myocardial infarction within 6 months before the Screening
   2. Unstable angina within 3 months before the Screening
   3. New York Heart Association class III or IV congestive heart failure
   4. History of sustained ventricular tachycardia, ventricular fibrillation, and/or Torsades de Pointes
   5. QT interval corrected by Fridericia's formula > 480 milliseconds
   6. History of Mobitz II second-degree or third-degree heart block without a permanent pacemaker in place
2. History of central nervous system (CNS) hemorrhage
3. Documented progressive disease (PD) during ibrutinib and/or acalabrutinib treatment.
4. Have received any anticancer therapy (other than immunotherapy) for CLL/SLL, WM, MCL, and MZL < 7 days before any Screening assessments are performed or any immunotherapy treatment, taken alone or as part of a chemoimmunotherapy regimen, < 4 weeks before any Screening assessments are performed
5. Requires ongoing need for corticosteroid treatment > 10 mg daily of prednisone or equivalent corticosteroid. Note: Systemic corticosteroids must be fully tapered off/discontinued ≥ 5 days before the first dose of study drug is administered.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2026-01-09 (Actual); Study Completion 2026-01-09 (Actual)

PRIMARY OUTCOMES:
Recurrence and change in severity of treatment-emergent Adverse Events (AEs) of interest. | 24 months

SECONDARY OUTCOMES:
Overall response as determined by investigator | 24 months
Progression free survival (PFS) as determined by investigator | 24 months
Patient reported outcomes as measured by EuroQol five dimension scale (EQ-5D) | 24 months
Patient reported outcomes as measured by European Organisation for Research and Treatment of Cancer (EORTC) | 24 months
Disease control rate as determined by investigator | 24 months

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Rocky Mountain Cancer Centers (Williams) Usor, Aurora, Colorado
  - Christiana Care, Newark, Delaware
  - Scri Florida Cancer Specialists South, Fort Myers, Florida
  - St Century Oncology, Jacksonville, Florida
  - Scri Florida Cancer Specialists North, St. Petersburg, Florida
  - Healthcare Research Network Iii, Llc, Flossmoor, Illinois
  - Minnesota Oncology Burnsville Clinic, Burnsville, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Summit Medical Group, Florham Park, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Clinical Research Alliance, Inc, Westbury, New York
  - Oncology Associates of Oregon Willamette Valley Cancer Center, Eugene, Oregon
  - St Lukes University Health Network, Fountain Hill, Pennsylvania
  - Abington Hematology Oncology Associates, Horsham, Pennsylvania
  - Tennessee Oncology, Pllc Nashville, Nashville, Tennessee
  - Texas Oncology Amarillo, Amarillo, Texas
  - Texas Oncology Tyler Longview, Austin, Texas
  - Baylor Research Institute, Dallas, Texas
  - Texas Oncology McAllen South Second Street, McAllen, Texas
  - Us Oncology Virginia Cancer Specialists, Pc, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical Oncology Associates, Spokane, Washington
  - Ssm Health Cancer Care Dean Medical Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/

REFERENCES:
- [Derived] Shadman M, Burke JM, Cultrera J, Yimer HA, Zafar SF, Misleh J, Rao SS, Farber CM, Cohen A, Yao H, Idoine A, An Q, Flinn IW, Sharman JP. Zanubrutinib is well tolerated and effective in patients with CLL/SLL intolerant of ibrutinib/acalabrutinib: updated results. Blood Adv. 2025 Aug 26;9(16):4100-4110. doi: 10.1182/bloodadvances.2024015493. PMID 40334067
- [Derived] Shadman M, Flinn IW, Levy MY, Porter RF, Burke JM, Zafar SF, Misleh J, Kingsley EC, Yimer HA, Freeman B, Rao SS, Chaudhry A, Tumula PK, Gandhi MD, Manda S, Chen DY, By K, Xu L, Liu Y, Crescenzo R, Idoine A, Zhang X, Cohen A, Huang J, Sharman JP. Zanubrutinib in patients with previously treated B-cell malignancies intolerant of previous Bruton tyrosine kinase inhibitors in the USA: a phase 2, open-label, single-arm study. Lancet Haematol. 2023 Jan;10(1):e35-e45. doi: 10.1016/S2352-3026(22)00320-9. Epub 2022 Nov 16. PMID 36400069